CLINICAL TRIAL: NCT03879356
Title: Supportive Measures in Treatment of Aluminum Phosphide Poisoning as a Trial to Reduce Mortality at Assiut University Hospital
Brief Title: Supportive Measures in Treatment of Aluminum Phosphide Poisoning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MKMAbdelrahim, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AluminumPhosphideAssiut
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Detection of Different Prognostic Factors and Their Relation With the Outcome; Using New Protocol to Prove the Role of N-acetyl Cysteine and Adequate Supportive Measures in Aluminum Phosphide Poisoning
Keywords: Aluminum phosphide; N-acetylcystein; Assiut; prognostic factors
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aluminum phosphide patients (Other): effect of N-acetyl cysteine and supportive measures in outcome of aluminum phosphide poisoning cases
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — effect of N-acetyl cysteine in Aluminum phosphide poisoning patients

SUMMARY:
Aluminum phosphide poisoning (ALP) is a global public health problem, and self-poisoning accounts for one-third of the world's suicide rate. In fact, in some parts of developing countries, pesticide poisoning causes more deaths than infection. ALP is very common in our government and the prognosis of the cases is usually so bad. Toxicity by ALP is caused by the liberation of phosphine gas, which causes cell hypoxia due to inhibition of oxidative phosphorylation leading to circulatory failure.

DETAILED DESCRIPTION:
Aluminum phosphide poisoning is a major problem, accounting for many Emergency Unit visits and hospitalization, the incidence of aluminum phosphide poisoning increasing in the last few years.

ALP is used as pesticides for many years to protect grains in stores and during its transportation. The availability of these tablets and their low cost make it an easy and common method of suicide in our country with the increasing incidence of social and financial problems that face the youth.

In management, the main objective is to provide effective oxygenation, ventilation, and circulation until phosphine is excreted. All patients of severe ALP poisoning require continuous invasive hemodynamic monitoring and early resuscitation with fluid and vasoactive agents. N- acetylcysteine as an antioxidant and cytoprotective agent reduces myocardial oxidative injury and increase survival time. Magnesium sulfate helps in scavenging free radicals through glutathione (GSH) recovery hence is effective as a parenteral antioxidant in this poisoning as well as has been tried for its general membrane stabilizing effect in cardiac cells .

Death after 24 hours occurs usually owing to shock, cardiac arrhythmia, metabolic acidosis, and acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All the cases with the primary diagnosis of Aluminum phosphide toxicity will be included in the study.
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients with a history of any chronic disease (renal and hepatic).
* Patients refuse to participate in the study.
* Aged less than 18 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
mortality rate comparison | 3 days
  comparison of mortality rate using the New protocol and previous mortality rate from archive records
hospital stay | 3 days
  number of days the patient stayed at hospital